CLINICAL TRIAL: NCT01058161
Title: High-Field MRI Characterization of Wrist and Hand Cartilage Abnormalities in Inflammatory and Chronic Rheumatisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-A01040-57; 2009 28 (Other: 2009 28)
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Abnormality; Inflammation; Rheumatism
Keywords: wrist and hand cartilage abnormalities in inflammatory and chronic rheumatisms
MeSH Terms: conditions — Congenital Abnormalities; Inflammation; Rheumatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Suspects or affected by rheumatoid polyarthritis (Other)
  Interventions: Other: high-field MRI (3 Teslas)
- stiffening spondylitis with axial and peripheral infringement (Other)
  Interventions: Other: high-field MRI (3 Teslas)
- polyarthralgies with or without arthritis (Other): Affected by connectivity with anti-nuclear antibody positive and / or specific antibodies, suffering of polyarthralgias with or without arthritis
  Interventions: Other: high-field MRI (3 Teslas)
- Healthy control (Other)
  Interventions: Other: high-field MRI (3 Teslas)
- not inflammatory control (Other): Presenting a degenerative osteoarthritis of the wrist traumatic comment, noticed radiologically, which will serve as not inflammatory control.
  Interventions: Other: high-field MRI (3 Teslas)

INTERVENTIONS:
Other: high-field MRI (3 Teslas) — high-field MRI (3 Teslas)
Other: high-field MRI (3 Teslas) — high-field MRI (3 Teslas)
  Arms: stiffening spondylitis with axial and peripheral infringement
Other: high-field MRI (3 Teslas) — high-field MRI (3 Teslas)
  Arms: polyarthralgies with or without arthritis
Other: high-field MRI (3 Teslas) — high-field MRI (3 Teslas)
  Arms: Healthy control; not inflammatory control

SUMMARY:
The present project aims at evaluating the diagnostic potential of high-field MRI (3 Teslas) for joint disease. At this field, given that isotropic image resolution of 400 microns can be obtained, one could expect an early detection of joint abnormalities. The additional aim of this project will be to develop a quantitative analyse of the corresponding high-resolution images.

ELIGIBILITY:
Inclusion Criteria:

* gp Suspects or affected by rheumatoid polyarthritis

  1. Morning articular Stiffness of at least 15 minutes.
  2. Arthalgias or Arthritises of at least three joints(articulations), among which those of the hand.
  3. Possible rheumatoid Presence of a factor(mailman) and\or Antibody anti peptides positive citrullinés.
  4. Typical possible radiological Hurts on the standard clichés(pictures) of the reached(affected) joints(articulations).
* gp Affected by stiffening spondylitis with axial and peripheral infringement :

  . Lumbago and steepness lumbar vertebra inflammatory. 2. Arthralgias and\or peripheral arthritises 3. Possible presence of an allèle HLA 4. Possible presence of a sacro-illite 5. Absence of the other rheumatic markers
* gp Affected by connectivity with anti-nuclear antibody positive and / or specific antibodies, suffering of polyarthralgias with or without arthritis
* gp Healthy control
* gp Presenting a degenerative osteoarthritis of the wrist traumatic comment, noticed radiologically, which will serve as not inflammatory control.

Exclusion Criteria:

* Claustrophobia,
* metallic foreign bodies,
* pacemakers The pregnant women,
* parturients or who breast-feed are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
can be obtained, one could expect an early detection of joint abnormalities | 24 months

SECONDARY OUTCOMES:
will be to develop a quantitative analyse of the corresponding high-resolution images. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: sandrine guis, PU PH, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France